CLINICAL TRIAL: NCT00472420
Title: An Open-label Study of the Effect of the Addition of MabThera to Standard Chemotherapy on Clinical Response in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: A Study of MabThera (Rituximab) Plus Standard Chemotherapy in Patients With Previously Untreated Mantle Cell Lymphoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20493
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: First line chemotherapy

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375mg/m2 iv every 3 weeks
Drug: First line chemotherapy — As prescribed

SUMMARY:
This single arm study will evaluate the benefit of adding MabThera to standard induction chemotherapy in patients with newly diagnosed mantle cell lymphoma. The safety and tolerability of a MabThera-containing first line regimen will also be assessed. All patients will receive MabThera (375mg/m2 iv) every 3 weeks for 8 cycles, in combination with standard chemotherapy. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* histologically-proven mantle cell lymphoma;
* previously untreated disease at stage II, III and IV, requiring therapy.

Exclusion Criteria:

* known hypersensitivity reaction to rituximab, or known anti-murine antibody reactivity or known hypersensitivity to murine antibodies;
* active malignancy other than mantle cell lymphoma within 5 years of start of study, with the exception of resected basal cell cancer, squamous cell cancer of the skin, or in situ cancer of the cervix;
* serious disorders interfering with full standard dosing chemotherapy;
* stage I disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-06-27 (Actual); Primary Completion 2011-05-25 (Actual); Study Completion 2011-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Hungary (7):
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Institute of Internal Medicine, Hematology, Debrecen
  - Petz Aladar Megyei Korhaz; Hematologia, Győr
  - Kaposi Mor Teaching Hospital, Dept of Internal Medicine/Hematology, Kaposvár
  - Miskolci Semmelweis Korhaz; Ii Belgyogyaszat, Miskolc
  - University of Szeged, II Dept of Internal Medicine, Szeged
  - Zala Megyei Korhaz; Ii. Belgyogyaszat, Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus (+) Chemotherapy: Participants received rituximab, 375 milligrams per square meter (mg/m^2), intravenously (IV), on Day 1 of Cycles 1-8 (21-day cycle). Participants also received 1 of the following chemotherapies: CHOP, Cycles 1-8: cyclophosphamide, 750 mg/m^2, IV, doxorubicin, 50 mg/m^2, IV, or epirubicin, 70 mg/m^2, IV, vincristine, 1.4 mg/m^2, IV, on Day 1 of Cycles 1-8, and methylprednisolone, 16 mg/d, IV or orally (PO), on Days 1-5. OR Hyper-CVAD/M-A, Cycles 1, 3, 5, and 7: cyclophosphamide, 300 mg/m^2, IV, every 12 hours (q12h) on Days 2-4; mesna, 600 mg/m^2, IV, 1 hour before the start of cyclophosphamide on Days 2-4; doxorubicin, 50 mg/m^2, IV, or epirubicin, 70 mg/m^2, IV, on Day 5; vincristine, 1.4 mg/m^2, IV, on Days 5 and 12; and dexamethasone, IV or PO, 40 mg/day on Days 2-5 and Days 12-15. Hyper-CVAD/M-A, Cycles 2, 4, 6, and 8: methotrexate, 200 mg/m^2, IV, followed by 800 mg/m^2, IV, on Day 2; cytarabine, 3000 mg/m^2, IV over 2 hours, q12h on Day 3 (2 doses) or Days 3-4 (4 doses).
Period: Induction Treatment Period
Arm/Group | Rituximab Plus (+) Chemotherapy
Started | 48
Completed | 32
Not Completed | 16
Not completed — Physician Decision | 9
Not completed — Adverse Event | 3
Not completed — Non-compliance | 1
Not completed — Death | 3
Period: Follow-up Period
Arm/Group | Rituximab Plus (+) Chemotherapy
Started | 32
Completed | 15
Not Completed | 17
Not completed — Death | 5
Not completed — Physician Decision | 9
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants who received at least 1 dose of study treatment.
Groups:
- Rituximab + Chemotherapy: Participants received rituximab, 375 mg/m^2, IV, on Day 1 of Cycles 1-8 (21-day cycle). Participants also received 1 of the following chemotherapies: CHOP, Cycles 1-8: cyclophosphamide, 750 mg/m^2, IV, doxorubicin, 50 mg/m^2, IV, or epirubicin, 70 mg/m^2, IV, vincristine, 1.4 mg/m^2, IV, on Day 1 of Cycles 1-8, and methylprednisolone, 16 mg/d, IV or PO, on Days 1-5. OR Hyper-CVAD/M-A, Cycles 1, 3, 5, and 7: cyclophosphamide, 300 mg/m^2, IV, q12h on Days 2-4; mesna, 600 mg/m^2, IV, 1 hour before the start of cyclophosphamide on Days 2-4; doxorubicin, 50 mg/m^2, IV, or epirubicin, 70 mg/m^2, IV, on Day 5; vincristine, 1.4 mg/m^2, IV, on Days 5 and 12; and dexamethasone, IV or PO, 40 mg/day on Days 2-5 and Days 12-15. Hyper-CVAD/M-A, Cycles 2, 4, 6, and 8: methotrexate, 200 mg/m^2, IV, followed by 800 mg/m^2, IV, on Day 2; cytarabine, 3000 mg/m^2, IV over 2 hours, q12h on Day 3 (2 doses) or Days 3-4 (4 doses).
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] — 47 participants were included in the calculation of age.
  years | 70.20 [44.46 to 82.31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Complete Remission (CR) (Including Unconfirmed CR [CR(u)]) or Partial Remission (PR)
Description: CR was defined by: a) disappearance of clinical/radiographic evidence of disease, disease-related symptoms, and biochemical abnormalities; b) decrease in lymph nodes (LNs) greater than (>) 1.5 centimeters (cm) in greatest transverse diameter (GTD) to less than (<) 1.5 cm, a decrease in LNs 1.1 - 1.5 cm to 1 cm or 75 percent (%) decrease in sum of the products of GTD (SPD); c) non-palpable spleen, decreased size of enlarged organs, and disappearance of nodules; and d) disappearance of bone marrow (BM) infiltrate. CR(u) was defined as fulfilling a) and c), above, with greater than or equal to (≥) 1 of the following: a) > 75% decrease in SPD of LNs > 1.5 cm, and > 75% decrease in SPD of previously confluent LNs; b) indeterminate BM, or c) confirmed CR. PR was defined by: a) 50% decrease in SPD of the 6 largest LNs; b) no increase in LNs, liver, or spleen size; c) ≥ 50% decrease in splenic and hepatic nodule SPDs; d) no measurable disease in other organs; and e) no new sites of disease.
Time Frame: Screening, Baseline (BL), every 21 days thereafter up to Week 27, every 3 months thereafter up to Month 24, Withdrawal Visit (4 weeks after discontinuation of study treatment)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 48
participants
  CR | 19
  PR | 8

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the median time, in months, from the date of study entry to disease progression, death due to mantle cell lymphoma, or last contact. Progressive disease (PD) was defined by: a) 50% increase from nadir in the SPD of any previously identified abnormal LN, or b) appearance of any new lesion during or at the end of treatment. The 95% confidence interval (CI) was estimated using Kaplan-Meier methodology.
Time Frame: Screening, BL, every 21 days thereafter up to Week 27, every 3 months thereafter up to Month 24, Withdrawal Visit (4 weeks after discontinuation of study treatment)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 48
months | 30.456 [19.011 to 41.901]

3. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the median time, in months, from the date of study entry disease progression, relapse, secondary malignancy, death or last contact. Relapse was defined by: a) appearance of any new lesion or a ≥ 50% increase in size of previously involved sites, or b) ≥ 50% increase in GTD of any previously identified LN >1 cm in short axis or in the SPD of more than one LN. The 95% CI was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 2
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 48
months | 40.049 [33.296 to 46.802]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded throughout the study up to 3 months after the last study drug administration.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis.
Arm/Group | Rituximab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 25/48
Other Adverse Events (participants affected / at risk) | 23/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=48)
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Septic shock (Infections and infestations) | 1
Pyrexia (General disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 6
Nausea (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Sinusitis (Infections and infestations) | 1
Pleurlopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Arrythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Tumour excision (Surgical and medical procedures) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Acute coronaria syndrome (Cardiac disorders) | 1
Disease recurrence (General disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Periproctal abscess (Infections and infestations) | 1
Urticaria, perioral tingling (Skin and subcutaneous tissue disorders) | 1
Heart injury (Cardiac disorders) | 1
Progression of pre-existing cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 4
Encephalomalacia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=48)
Diarrhoea infectious (Gastrointestinal disorders) | 1
Bacteremia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Herpes zoster (Infections and infestations) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 5
Pancytopenia (Blood and lymphatic system disorders) | 2
Pruritus cutaneous (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Toxicoderma (Skin and subcutaneous tissue disorders) | 1
Helicobacter test positive (Infections and infestations) | 1
Chills (General disorders) | 4
Pyrexia (General disorders) | 3
Chilliness (General disorders) | 1
Pain (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 2
Oral thrush (Infections and infestations) | 1
Prostatitis (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes labialis (Infections and infestations) | 1
Bone marrow toxicity (Blood and lymphatic system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Ulcus corneae (Eye disorders) | 1
Carotid sinus syndrome (Cardiac disorders) | 1
Choking sensation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.